CLINICAL TRIAL: NCT01696214
Title: SAPS:Smoking Asthmatics Pilot Study:
Brief Title: A Pilot Study to Determine the Feasibility and Utility of Implementing of the Full Scale TOM Trial
Acronym: SAPS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Joe Ramsdell, Medical Doctor, University of California, San Diego
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: ARCTC-09; IR34HL109482-01A1 (Other Grant/Funding Number: National Heart, Lung, and Blood Institute (NHLBI))
Record Dates: First submitted 2012-06-25; First posted 2012-09-28 (Estimated); Results first posted 2016-10-12 (Estimated); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Asthma
Keywords: asthma,smokers
MeSH Terms: conditions — Asthma | interventions — Fluticasone; Salmeterol Xinafoate; montelukast; Theophylline; Ipratropium

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Ipratropium (Placebo Comparator): Participants will continue fluticasone 100 mg/salmeterol 50 mg once a day and be assigned to a 24 week treatment of ipratropium 2.5 mL, 0.02% 3 times daily via mini nebulizer with placebo theophylline and placebo montelukast.
  Interventions: Drug: ipratropium
- Theophylline (Placebo Comparator): Participants will continue fluticasone 100 mg/salmeterol 50 mg once a day and will be assigned to theophylline 400 mg once a day for 24 weeks with placebo ipratropium and placebo montelukast.
  Interventions: Drug: Theophylline 400 mg
- Montelukast (Placebo Comparator): Participants will continue fluticasone 100 mg/salmeterol 50 mg once a day and will be assigned to montelukast 10 mg once a day for 24 weeks with placebo theophylline and placebo ipratropium.
  Interventions: Drug: Montelukast 10mg
- fluticasone 250 mg/salmeterol 50mg (Placebo Comparator): Participants will be assigned to inhaled fluticasone 250/salmeterol 50 twice a day for 24 weeks with placebo theophylline, placebo ipratropium, and placebo montelukast.
  Interventions: Drug: Fluticasone 250 mg/salmeterol 50 mg

INTERVENTIONS:
Drug: Fluticasone 250 mg/salmeterol 50 mg — Drug: Fluticasone 250 mg/salmeterol 50 mg Participants will be assigned to a 24 week treatment with inhaled fluticasone/salmeterol or matching placebo
  Other Names: Advair(fluticasone/salmeterol)250/50
  Arms: fluticasone 250 mg/salmeterol 50mg
Drug: Montelukast 10mg — Participants will be assigned to montelukast once a day for 24 weeks.
  Other Names: Singulair
  Arms: Montelukast
Drug: Theophylline 400 mg — Participants will be assigned to theophylline once a day for 24 weeks
  Arms: Theophylline
Drug: ipratropium — Participants will be assigned to ipratropium 2.5 mL of 0.02% solution via mini nebulizer 3 times a day day for 24 weeks.
  Other Names: Atrovent
  Arms: Ipratropium

SUMMARY:
The primary aim of the pilot (SAPS) protocol is to determine the feasibility and utility of implementing the provisional design of the full scale TOM trial (e.g., the six month treatment period, the impact of the smoking cessation intervention).

There is no active hypothesis for the Vanguard Protocol.

DETAILED DESCRIPTION:
The protocol is a small scale pilot of the full-scale TOM trial, and it will utilize a placebo design and incorporates 4 treatment arms. In the Vanguard Protocol all participants are to complete a 4 week run-in with Advair 100/50, followed by randomization to 1 of 4 arms of study treatment. The 4 drug treatment combinations are (2 inhalers, 2 pills):

* Advair 250/50, Placebo, Placebo, Placebo
* Advair 100/50 and montelukast, Placebo, Placebo
* Advair 100/50 and theophylline, Placebo, Placebo
* Advair 100/50 and ipratropium, Placebo, Placebo The 24 week treatment phase will be followed by a 4 week washout period on Advair 100/50. There is no crossover.

ELIGIBILITY:
Inclusion Criteria:

* Gender and Age:
* Males and females, ages 18- 50

Current Smoker:

* Smoke at least 5 cigarettes per day for at least 5 years
* Positive urine cotinine test

Asthma:

* Physician diagnosed asthma
* Symptomatic, as evidenced by

  * Use of SABA two or more times per week for relief of asthma symptoms, or
  * One or more nocturnal awakenings per week for asthma symptoms ACRC - SC MEETING - 19 MAY 2012 SAPS │ 25 Confidential, not for attribution or citation.
* Pre-BD FEV1 greater than or equal to 40% predicted
* Asthma diagnosis confirmed by either

  * albuterol reversibility of FEV1 by 12% or more, or
  * 20% fall in FEV1 at 8mg or less of methacholine
* If over age 45, a DLco greater than 80% predicted
* Females of childbearing potential: not pregnant, not lactating and agree to practice an adequate birth control method (abstinence, combination barrier and spermicide, or hormonal) for the duration of the study.

Exclusion Criteria:

* Diagnosis of COPD or emphysema
* Other major chronic illnesses in the opinion of the investigator that might interfere with the study:

  - e.g. including but not limited to uncontrolled diabetes, uncontrolled HIV infection or other immune system disorder, hyperthyroidism, seizure disorders, renal failure, liver disease, non-skin cancer, unstable psychiatric illness.
* Recent active substance abuse (in past 6 months)
* Lung disease other than asthma including COPD, bronchiectasis, sarcoidosis, or other significant lung disease
* Unstable cardiac disease (decompensated CHF, unstable angina, recent MI, atrial fibrillation, supraventricular or ventricular tachycardia, congenital heart disease, or severe uncontrolled hypertension).
* High risk of near fatal or fatal asthma as defined by the following 1-3

  * ICU admission of asthma in the past year
  * more than 2 hospitalizations for asthma in the previous year
  * more than 3 ED visits for asthma in the previous year
  * intubation or ICU admission for asthma in the past 2 years
  * use of more than 2 canisters of inhaled short-acting beta2-agonist in past month
* Acute asthma exacerbation in the past 4 weeks (treatment with systemic corticosteroids)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2012-10; Primary Completion 2015-05 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joe Ramsdell, MD, Principal Investigator — UCSD
Locations (1):
- Airway Research & Clinical Trials Center, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: Yes
results will be presented been publication four-minute meetings

RESULTS

PARTICIPANT FLOW:
Groups:
- Ipratropium: Participants will continue fluticasone 100 mg/salmeterol 50 mg once a day and be assigned to a 24 week treatment of ipratropium 0.02% solution, 2.5 ml via mini nebulizer for 24 weeks with placebo theophylline and placebo montelukast.
  Ipratropium: Participants will be assigned to ipratropium 0.02% solution, 2.5 ml via mini nebulizer 3 times
- Theophylline: Participants will continue fluticasone 100 mg/salmeterol 50 mg once a day and will be assigned to theophylline 400 mg once a day for 24 weeks with placebo ipratropium and placebo montelukast.
  Theophylline: Participants will be assigned to theophylline 400 mg once a day for 24 weeks
- Montelukast: Participants will continue fluticasone 100 mg/salmeterol 50 mg once a day and will be assigned to montelukast 10 mg once a day for 24 weeks with placebo theophylline and placebo ipratropium.
  Montelukast 10mg: Participants will be assigned to montelukast 10 mg once a day for 24 weeks.
- Fluticasone 250 mg/Salmeterol 50mg: Participants will be assigned to inhaled fluticasone 250 mg/salmeterol 50 mg twice a day for 24 weeks with placebo theophylline, placebo ipratropium, and placebo montelukast.
  Fluticasone 250 mg/salmeterol 50 mg:
  Participants will be assigned to a 24 week treatment with inhaled fluticasone 250 mg /salmeterol 50
Period: Overall Study
Arm/Group | Ipratropium | Theophylline | Montelukast | Fluticasone 250 mg/Salmeterol 50mg
Started | 5 | 5 | 5 | 5
Completed | 4 | 5 | 5 | 5
Not Completed | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: smoking asthmatics
Groups:
- Ipratropium: Participants will continue fluticasone 100 mg/salmeterol 50 mg once a day and be assigned to a 24 week treatment of ipratropium 0.02% solution, 2.5 ml via mini nebulizer for 24 weeks with placebo theophylline and montelukast.
  Ipratropium: Participants will be assigned to ipratropium 0.02% solution, 2.5 ml via mini nebulizer 3 times
- Theophylline: Participants will continue fluticasone 100 mg/salmeterol 50 mg once a day and will be assigned to theophylline 300 mg once a day for 24 weeks with placebo tiotroprium and montelukast.
  Theophylline: Participants will be assigned to theophylline 300 mg once a day for 24 weeks
- Montelukast: Participants will continue fluticasone 100 mg/salmeterol 50 mg once a day and will be assigned to montelukast 10 mg once a day for 24 weeks with placebo theophylline and tiotroprium.
  Montelukast 10mg: Participants will be assigned to montelukast 10 mg once a day for 24 weeks.
- Fluticasone 250 mg/Salmeterol 50mg: Participants will be assigned to inhaled fluticasone 250 mg/salmeterol 50 mg twice a day for 24 weeks with placebo theophylline, tiotroprium, and montelukast.
  Fluticasone 250 mg/salmeterol 50 mg:
  Participants will be assigned to a 24 week treatment with inhaled fluticasone 250 mg /salmeterol 50
- Total: Total of all reporting groups
Arm/Group | Ipratropium | Theophylline | Montelukast | Fluticasone 250 mg/Salmeterol 50mg | Total
Number analyzed (Participants) | 4 | 5 | 5 | 5 | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 5 | 5 | 5 | 19
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 49 [42 to 50] | 48 [44 to 50] | 39 [28 to 50] | 28 [26 to 50] | 41 [26 to 50]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 3 | 1 | 10
  Male | 0 | 3 | 2 | 4 | 9
Region of Enrollment [Number; unit: participants]
  United States | 4 | 5 | 5 | 5 | 19

OUTCOME MEASURES:

1. Primary Outcome: Asthma Control Test
Description: The primary symptomatic measure, the Asthma Control Test (ACT), has been shown to be valid for measuring poor asthma control in asthmatic children and non-smoking adults. The ACT is a tool developed by Nathan and collaborators a decade ago for evaluating asthma control. It consists of five questions with five possible answers each. A maximum score of 25 points indicates complete asthma control. A score between 20 and 24 represents partially controlled asthma, while a score 19 or below indicates poorly controlled asthma and a score <16 indicates uncontrolled asthma. The minimally important clinical difference has been determined to be 3.
Time Frame: Outcome measure was assessed at the initial visit, at randomization following a wash-in period of 1 month, monthly for 24 weeks and at follow-up visit 1 month off study drug. Median scores over the 24 weeks of treatment were compared.
Measure: Median (Full Range); unit: units on a scale
Groups:
- Ipratropium: Participants will continue fluticasone 100 mg/salmeterol 50 mg once a day and be assigned to a 24 week treatment of ipratropium 2.5 mL, 0.02% 3 times daily via mini nebulizer with placebo theophylline and montelukast.
  ipratropium: Participants will be assigned to ipratropium 2.5 mL of 0.02% solution via mini nebulizer 3 times a day day for 24 weeks.
- Theophylline: Participants will continue fluticasone 100 mg/salmeterol 50 mg once a day and will be assigned to theophylline 400 mg once a day for 24 weeks with placebo ipratropium and montelukast.
  Theophylline 400 mg: Participants will be assigned to Theophylline once a day for 24 weeks
- Montelukast: Participants will continue fluticasone 100 mg/salmeterol 50 mg once a day and will be assigned to montelukast 10 mg once a day for 24 weeks with placebo theophylline and ipratropium.
  Montelukast 10mg: Participants will be assigned to Leukotriene receptor antagonist once a day for 24 weeks.
- Fluticasone 250 mg/Salmeterol 50mg: Participants will be assigned to inhaled fluticasone 250/salmeterol 50 twice a day for 24 weeks with placebo theophylline, ipratropium, and montelukast.
  Fluticasone 250 mg/salmeterol 50 mg: Drug: Fluticasone 250 mg/salmeterol 50 mg Participants will be assigned to a 24 week treatment with inhaled fluticasone/salmeterol or matching placebo
Arm/Group | Ipratropium | Theophylline | Montelukast | Fluticasone 250 mg/Salmeterol 50mg
Number analyzed (Participants) | 4 | 5 | 5 | 5
units on a scale | 17.5 [13 to 19] | 13 [7 to 19] | 12 [9 to 15] | 10 [5 to 13]

2. Secondary Outcome: The Asthma Symptom Utility Index (ASUI)
Description: The Asthma Symptom Utility Index (ASUI), an important secondary outcome in the proposed full-scale TOM Trial, has also been shown to be useful in tracking the frequency and severity of asthma-related symptoms in non-smoking asthmatics. ASUI is a brief, interviewer-administered, patient preference-based scale assessing frequency and severity of selected asthma-related symptoms and treatment side effects. 11 items are reviewed, with 2-week recall to assess four symptoms (cough, wheeze, shortness of breath, and awakening at night) and medication side-effects each on two dimensions (frequency and severity). 4-point Likert scale is used to assess frequency (not at all, 1 to 3 days, 4 to 7 days, and 8 to 14 days) and severity (not applicable, mild, moderate and severe). Scores range from 0 (worst possible symptoms) to 1 (no symptoms). The change between two time points, initial visit and after 24 weeks of treatment, is reported. The median value is reported with the standard deviation.
Time Frame: Outcome measure was assessed at the initial visit, at randomization following a wash-in period of 1 month, monthly for 24 weeks and a follow-up visit 1 month off study drug. Median scores, change from initial visit and end of treatment, were compared
Measure: Median (Standard Deviation); unit: units on a scale
Arm/Group | Ipratropium | Theophylline | Montelukast | Fluticasone 250 mg/Salmeterol 50mg
Number analyzed (Participants) | 4 | 5 | 5 | 5
units on a scale | 0.16 (0.07) | 0.24 (0.20) | 0.14 (0.15) | 0.13 (0.18)

3. Secondary Outcome: Percent (%) Perdicted FEV1 Changes
Description: Physiologic measures of % predicted FEV1
Time Frame: Outcome measure was assessed at the initial visit, at randomization following a wash-in period of 1 month, monthly for 24 weeks. Median scores over the 24 weeks of treatment were compared
Measure: Median (Standard Deviation); unit: percent predicted FEV1
Arm/Group | Ipratropium | Theophylline | Montelukast | Fluticasone 250 mg/Salmeterol 50mg
Number analyzed (Participants) | 4 | 5 | 5 | 5
percent predicted FEV1 | -1.62 (7.89) | 4.73 (7.72) | 0.87 (10.57) | -5.71 (5.24)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Ipratropium | Theophylline | Montelukast | Fluticasone 250 mg/Salmeterol 50mg
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/5 | 1/5 | 0/5
Other Adverse Events (participants affected / at risk) | 4/5 | 5/5 | 5/5 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ipratropium (N=4) | Theophylline (N=5) | Montelukast (N=5) | Fluticasone 250 mg/Salmeterol 50mg (N=5)
asthma exacerbation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Participant hospitalized overnight with asthma exacerbation. Study drug stopped while overnight hospitalization and continued with randomized study drug and completed double blind portion of study.
death (Social circumstances) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Participant in the run-out phase with open label Advair 100/50 and was found dead. Autopsy found cause of that to be due to Phencyclidine and Cocaine Toxicity
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ipratropium (N=5) | Theophylline (N=5) | Montelukast (N=5) | Fluticasone 250 mg/Salmeterol 50mg (N=5)
migraine headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — migraine headache
viral infection (Infections and infestations) | 4 (4) | 1 (1) | 1 (1) | 3 (3) — self-limiting viral infection
back pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 1 (1) | 0 (0) — transient back pain
drowsiness (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — transient drowsiness
rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — transient rash
motor vehicle accident (Social circumstances) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — motor vehicle accident with no serious injury
dry mouth (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — transient dry mouth
chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — transient chest wall discomfort
urinary tract infection (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — treated urinary tract infection with no recurrence
nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) — transient nausea
diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — transient diarrhea
tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) — transient tachycardia
headache (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) — musculoskeletal headache
edema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — mild transient edema
skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — stable keratosis
swollen hand (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — transient swollen hand
constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — transient constipation
sprained finger (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — sprained finger, recovered without difficulty
pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — transient lower extremity itching
iritis (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — transient viral

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No